CLINICAL TRIAL: NCT07125222
Title: Use of Gocovri to Improve Disability Due to Radiation Encephalopathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Supernus Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-10026601
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Radiation Encephalopathy
MeSH Terms: interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gocovri (extended-release amantidine) (Experimental)
  Interventions: Drug: Gocovri (extended-release amantidine)

INTERVENTIONS:
Drug: Gocovri (extended-release amantidine) — Gocovri is extended release formulation of amantidine. Starting on Day 1, patients will start Gocovri 137mg daily. If there is no dose-limited event after 28 days, the dose will be increased to 274mg daily which will become the new standard dose for the remaining 20 weeks of the patient's participation in the study.

SUMMARY:
A study to assess the effect of Gocovri (extended-release amantidine) to improve disability as assessed by the disability rating scale (DRS) and cognition as assessed by the Montreal Cognitive Assessment (MoCA) test in patients with radiation encephalopathy.

DETAILED DESCRIPTION:
This is a prospective study to assess the effect of Gocovri (extended-release amantidine) on disability and cognition in patients with radiation encephalopathy. Patients with radiation encephalopathy will be seen in the office, and both clinical and short structured neuropsychological assessments will be collected longitudinally as medication adjustments are performed over time. The investigators will also measure functional glutamate activity in these subjects through use of F-FPEB PET/CT, which identifies mGluR5 expression in the brain. This imaging tracer serves as a surrogate for neurodegeneration in other conditions, such as Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age.
* Individuals with caregivers who are able to complete survey assessments for this study.
* Prior brain radiation treatment.
* Evidence of moderate-severe confluent white matter hyperintensity on MRI brain scan as judged by neuroradiology impression 0-5 years prior to enrollment.
* DRS > 6
* The effects of Gocovri on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (e.g. hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; female subjects will be required to demonstrate a negative urine pregnancy test prior to study entry and subjects who are lactating should be excluded.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Patients with growing brain lesions or those requiring escalating doses of tumor-directed treatment..
* Patients requiring doses of Dexamethasone higher than 4 mg or escalating doses of Dexamethasone
* Patients taking Amantadine or with prior usage of Amantadine.
* Patients taking other dopaminergic, GABAergic, glutamatergic, or noradrenergic drugs.
* Patients with a history of suicidality and depression.
* Patients with end stage renal disease (creatinine clearance less than 15 mL/min/1.73 m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in the level of disability as measured by the Disability Rating Scale(DRS) | Baseline - 24 weeks.
  The Disability Rating Scale (DRS) is a tool used to evaluate impairment, disability and handicap caused by brain injury. Scores range from 0 (No disability) to a maximum of 29 (indicating an extreme vegetative state).

SECONDARY OUTCOMES:
Change in cognition based on the MoCA test. | Baseline - 24 weeks.
  The Montreal Cognitive Assessment (MoCA) is a brief screening tool to assess cognitive function and identify potential cognitive impairment. A score of 26-30 is considered normal, 18-25 as mild cognitive impairment, 10-17 as moderate cognitive impairment and below 10 as severe cognitive impairment.
Change in 18F-FPEB avidity on PET/CT. | Baseline - 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv S Magge, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided